CLINICAL TRIAL: NCT00141479
Title: A Single-center Safety and Tolerability Study to Evaluate the Impact of Treatment Interruption on Re-initiation of Bifeprunox in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: To Evaluate the Impact of Treatment Interruption on Re-initiation of Bifeprunox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: H. Lundbeck A/S (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: S154.2.013
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2006-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Treatment interruption on reinitiation; Schizophrenia; Schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — bifeprunox

INTERVENTIONS:
Drug: Bifeprunox

SUMMARY:
The purpose of this study is to investigate a safe treatment interruption interval(s) for re-initiation of bifeprunox at a therapeutic dose. The study duration is approximately 7 to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia or Schizoaffective disorder
* 18-55 years

Exclusion Criteria:

* Subjects who are acutely psychotic
* Subjects with current Axis I primary psychiatric diagnosis other than schizophrenia
* Subjects at significant risk of suicide
* Subjects with a seizure disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Wichita, Kansas, United States